CLINICAL TRIAL: NCT05713643
Title: Erector Spinae Plane Block Versus Paravertebral Block Versus Quadratus Lumborum Block on Postoperative Analgesia After Pelvi-ureteric Surgeries: A Randomized Double-Blinded, Non-inferiority Trial
Brief Title: ESPB vs PVB vs QLB After Pelvi-ureteric Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 50-12-12
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Erector Spinae Plane Block; Paravertebral Block; Quadratus Lumborum Block; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESPB group (Active Comparator)
  Interventions: Procedure: ESPB Technique
- TPVB group (Active Comparator)
  Interventions: Procedure: TPVB Technique
- QLB group (Active Comparator)
  Interventions: Procedure: QLB Technique

INTERVENTIONS:
Procedure: ESPB Technique — The patient will be in sitting position. The probe will be positioned with longitudinal alignment, 3 cm lateral to the spinous procedure of T8 to obtain a parasagittal view. An echogenic needle will be introduced from the caudal end of the probe and advanced in-plane direction until the needle tip hit the tip of the transverse process. Bupivacaine will be afterwards injected into the erector spinae plane block. Linear spread cranially and caudally below the muscle upon injection will be visualized on the US screen indicating successful block.
  Arms: ESPB group
Procedure: TPVB Technique — The patient will be in sitting position. The probe will be positioned with longitudinal alignment, 3 cm lateral and parallel to 8th spinous process till transverse process, superior costotransverse ligament, and pleura will be visualized then lateral tilt of the probe was done for better visualization of the PVS between the superior costotransverse ligament and the pleura. An echogenic needle was introduced at caudal end of transducer using the in-plane technique till piercing the superior costotransverse ligament . Bupivacaine will be injected into the PVS with downward displacement of the pleura indicating a successful block.
  Arms: TPVB group
Procedure: QLB Technique — The patient will be in lateral position. The probe will be placed above the iliac crest. The Petit's triangle will be identified. The three abdominal muscles (i.e., the external oblique, internal oblique and transversus abdominus muscles) will be detected. Both the external oblique and internal oblique muscles will be followed posteriorly until the layers of the thoracolumbar fascia appear as a bright hyperechogenic line. The quadratus lumborum muscle appears below to the latissimus dorsi muscle. While performing the quadratus lumborum block, "Shamrock sign" is identified; the transverse process of L4 appears as a stem whereas the three muscles psoas muscle, quadratus lumborum muscle and erector spinae appear as the leaves. A 22G (50mm) needle was inserted using an in-plane technique along the posterior edge of the ultrasound probe in the anteromedial direction. The needle tip was placed between the quadratus lumborum muscle and the Erector spinae muscle.
  Arms: QLB group

SUMMARY:
The aim of this study is to compare the analgesic efficacy of erector spinae plane block versus thoracic paravertebral block versus quadratus lumborum block on postoperative analgesia after pelvi-ureteric surgeries.

DETAILED DESCRIPTION:
Opioid-based analgesia plays a significant role in the control of postsurgical pain; however, use of opioid may lead to significant side effects (e.g., nausea and vomiting) and adverse events (e.g. respiratory depression), which may be associated with significantly longer hospital stays and higher hospital costs in the postsurgical setting .

Thoracic paravertebral block (TPVB) is a classic trunk block with definite analgesic effect for both somatic and visceral pain.

Quadratus Lumborum block (QLB) is a widely used regional anesthesia technique as well. It has been used for reducing postoperative pain after cesarean section, laparotomy or laparoscopic procedure and hip surgery.

Erector spinae plane block (ESPB) is a novel inter-fascial plane block first introduced by Forero et al. in 2016 , providing wide-ranging analgesia in lung surgery, laparoscopy, mastectomy, and pediatric surgery. The proposed mechanism of ESPB is that distribution of local anesthetic solution spreads into the para-vertebral space and epidural space, which then blocks the dorsal, ventral, and traffic branches of spinal nerve.

ESPB, TPVB and QLB III have been shown to improve analgesic outcome after urological surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Both genders
* American Society of Anesthesiologists (ASA) physical status I-III
* Undergoing elective pelvi-ureteric surgeries.

Exclusion Criteria:

* Body Mass Index > 30 kg/m2.
* Contraindication of deep nerve block such as allergic to anesthetic drug, coagulation disorder, and infection at the injection site.
* Chronic opioids dependence or chronic pain over 3 months.
* Use of medication such as gabapentin-pregabalin could affect pain perception.
* Unable to communicate preoperatively due to severe dementia, language barrier, or neuropsychiatric disorder.
* Unable to perform nerve block procedure due to difficult anatomy through ultrasound scan.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
The total postoperative morphine consumption | 48 hours postoperatively
  Total amount of rescue analgesic in the first 48 hours postoperative will be measured.

SECONDARY OUTCOMES:
Access post-operative pain scores | 48 hours Postoperatively
  Postoperative pain will be accessed using Numeric Rating Scale which ranges from 0 to 10 points, with 0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Access time of first analgesic | 48 hours Postoperatively
  The time to first request of rescue analgesia will be recorded
Patients' satisfaction after surgery. | 48 hours Postoperatively
  The degree of patient satisfaction will be assessed on a 5-point scale: (0= extremely dissatisfied, 1= unsatisfied, 2= neither satisfied nor unsatisfied, 3= satisfied), 4= extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Fouad Algyar, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: One year after the end of the study